CLINICAL TRIAL: NCT02143245
Title: Diagnostic Accuracy of Synovial Biopsy for Implant-Related Shoulder Infections
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140167-01H
Record Dates: First submitted 2014-04-17; First posted 2014-05-21 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Total Shoulder Arthroplasty
Keywords: Shoulder Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Revision Population (Other): The study population is both men and women who have had previous shoulder surgery with symptoms suggestive of deep infection. These include the presence of pain, stiffness, and radiologic signs of infection including implant lucencies or migration.
  Patients in this population will undergo a synovial biopsy, in addition to undergoing an open tissue biopsy at the time of their procedure. Diagnostic accuracy will be compared, and all participants will be tracked over time.
  Interventions: Diagnostic Test: Synovial Biopsy; Diagnostic Test: Open Tissue Biopsy

INTERVENTIONS:
Diagnostic Test: Synovial Biopsy — Synovial biopsy is a procedure using a guided needle, where 6 to 8 small tissue samples with be extracted from the shoulder using an x-ray guided needle.
Diagnostic Test: Open Tissue Biopsy — During the standard of care revision surgery, 6 to 8 small tissue samples will be taken in order to test for infection. This is standard of care treatment. As part of this study, an additional 1 to 2 samples of tissue would be taken in order to develop a test to determine more precisely what type of infection there may be.

SUMMARY:
The purpose of this study is to determine the efficacy of retrieving tissue samples via an x-ray guided needle that is inserted into the infected tissue in the shoulder. The procedure using the guided needle is called a synovial biopsy versus an open tissue biopsy, which is done at the time of surgery. By doing the synovial biopsy prior to a revision surgery, the investigators hope to avoid more invasive intervention if it is not needed. Some patients may appear to have an infection but once the biopsy is taken and the results are read, there may not be an infection and therefore no need for a revision surgery.

DETAILED DESCRIPTION:
The primary research objective is to assess the diagnostic accuracy of percutaneous synovial biopsy for detection of implant-related intra-articular shoulder infections (IISI).

The secondary objectives are to document the frequency of pain associated with shoulder synovial biopsy and to determine the correlation and agreement of several indices of infection as a means of providing preliminary evidence toward a clinical decision rule to rule in or rule out the diagnosis of implant-related intra-articular shoulder infection.

The third objective is to determine the rates of (re)infection, functional outcomes, and quality of life, over a two year follow up period following revision surgery.

The fourth objective is to determine whether an association exists between the biopsy location within the joint and relative yield and positive culture rates.

The fifth objective is to identify, develop, and validate tissue-specific biomarkers for the detection of IISI.

It is our hypothesis that synovial biopsy is valid tool for use in the diagnosis of shoulder arthroplasty and fracture implant related infections.

ELIGIBILITY:
Inclusion Criteria:

1. Previous shoulder surgery including hemiarthroplasty, total shoulder arthroplasty or reverse total shoulder arthroplasty, or internal fixation for shoulder fractures
2. Suspicion of infection, including acute fever and complaints of pain and/or stiffness post operatively
3. Revision shoulder surgery for patients described in (1)
4. Provide consent

Exclusion Criteria:

1. signs or symptoms of bacteremia or sepsis requiring urgent treatment, which would preclude the possibility of synovial biopsy
2. Unable to speak or read English/French
3. Psychiatric illness that precludes informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Synovial Biopsy (test diagnostic) and Open Biopsy (reference standard) | Pre-operatively.
  To assess the diagnostic accuracy of percutaneous synovial biopsy (test procedure) for detection of implant-related intraarticular shoulder infections (IISI), in comparison to direct macroscopic synovial biopsy, from either arthroscopic or open procedures (the reference standard).
  To address the primary objective, standard diagnostic accuracy statistics (sensitivity, specificity, positive predictive value, negative predictive value, likelihood ratio) will be derived, comparing lab results from percutaneous synovial biopsy specimen collection to those of the reference standard test (open/arthroscopic).

SECONDARY OUTCOMES:
Reported Pain | 24-hours after biopsy.
  Using a visual analog scale, participants will rank their pain level 24-hours after the synovial biopsy. 0 indicating no pain, and 10 indicating the worst pain. A higher score indicates a worse outcome.

OTHER OUTCOMES:
Rates of Re-Infection | Post-Operatively up to 5 years.
  Participants will be monitored for re-infection after their revision surgery for 5-years. Higher incidences of infection indicate a worse outcome.
Constant Score | Post-operatively up to 5-years.
  The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points.The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).
Western Ontario Osteoarthritis of the Shoulder (WOOS) | Post-operatively up to 5-years.
  The Western Ontario Osteoarthritis of the Shoulder Index (WOOS) is a disease specific evaluation, proven to be an accurate and valid assessment of function after shoulder replacement. The WOOS is a patient-reported measure, 19-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome.
American Shoulder and Elbow Surgeons (ASES) | Post-operatively up to 5-years.
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
EQ-5D-5L | Post-operatively up to 5-years.
  The EQ-5D-5L quality of life questionnaire is a brief, easy to administer generic health status questionnaire, consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (each question rated 1-5), lower scores indicate better outcome. It also includes a visual analogue scale for recording an individual's rating of their current health-related quality of life (scale 0 to 100), where a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — The Ottawa Hospital
Locations (4):
- Canada (4):
  - St. Joseph's Health Care London, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Sacré-Coeur Hospital of Montreal, Montreal, Quebec